CLINICAL TRIAL: NCT00347087
Title: Effect of the Angiotensin II Receptor Antagonist Irbesartan on Insulin Sensitivity and Metabolic Profile in Patients With Chronic Heart Failure
Brief Title: Effect of Irbesartan on Insulin Sensitivity in Chronic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRIS HF 7/04
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Chronic Heart Failure
Keywords: Insulin sensitivity; chronic heart failure; metabolism
MeSH Terms: conditions — Insulin Resistance | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Irbesartan — up-titration over 4 weeks to target dose 300 mg od

SUMMARY:
To test whether treatment with the angiotensin II receptor antagonist Irbesartan improves insulin sensitivity and metabolic profile in patients with chronic heart failure.

DETAILED DESCRIPTION:
In CHF impaired insulin sensitivity is a common finding characterised by elevated fasting insulin levels and impaired effectiveness of insulin to utilise glucose in peripheral tissues, mainly in skeletal muscle tissue. Additionally, impaired insulin sensitivity, i.e. insulin resistance, progresses in parallel to severity of CHF and relates to major clinical symptoms such as reduced exercise capacity and muscle fatigue. In survival analyses, insulin resistance is a significant predictor of mortality, independently of and additionally to other established prognostic markers such as age, NYHA class, peak oxygen consumption, or LVEF. These findings indicate that insulin resistance is involved in CHF pathophysiology. Importantly, insulin resistance in CHF occurs independently of ischemic etiology. In ischaemic heart disease, however, insulin resistance as part of the metabolic syndrome is also an important prerequisite for the development of arteriosclerosis. Accordingly insulin resistance was found worst in CHF patients with ischemic etiology compared to patients with CHF due to dilated cardiomyopathy and those with ischaemic heart disease without heart failure. On the basis of these findings we hypothesise that therapeutically improving insulin sensitivity may have additional beneficial effects on energy utilisation and therefore improve clinical symptoms such as reduced exercise capacity and muscle fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. ambulatory patients with symptomatic chronic heart failure (NAHY II-IV)
2. ischemic etiology
3. LVEF ≤ 45%
4. standard medical treatment for CHF (such as diuretics, beta blockers, ACE inhibitors, aspirin or warfarin). Patients should be treated with ACI inhibitor for at least 12 months prior to enrolment into the study. Patients should not be treated with angiotensin II receptor antagonists during the study other than the trial medication. Further medical treatment such as spironolactone, amiodarone and others are allowed if the patient is on a stable dose at the beginning of the trial. Dosages should be kept stable during the trial except adjustment is judged necessary for clinical reason.
5. Patient should be hospitalised due to deterioration of the cardiac disease at least once in the last 12 months under ACE-I therapy.
6. age > 21 years
7. informed consent

Exclusion Criteria:

1. hospitalisation with intervention within 2 weeks of intended randomisation
2. unstable IHD or Myocardial infarction < 2 months
3. open diagnosed diabetes mellitus / antidiabetic treatment with insulin, metformin, sulfonylurea, glinides
4. COPD treated with steroids

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity assessment using intravenous glucose tolerance testing | 3 months

SECONDARY OUTCOMES:
Assessment of body composition using dual energy x-ray absorptiometry | 3 months
Assessment of exercise capacity on a treadmill including respiratory gas analysis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Doehner, MD, PhD, Principal Investigator — Applied Cachexia Research, Cardiology, Charite, Campus Virchow Klinikum
Locations (1):
- Applied Cachexia Research, Cardiology Dept. Charite Medical School, Virchow Klinikum, Berlin, Germany

REFERENCES:
- [Derived] Doehner W, Todorovic J, Kennecke C, Rauchhaus M, Sandek A, Lainscak M, van Linthout S, Tschope C, von Haehling S, Anker SD. Improved insulin sensitivity by the angiotensin receptor antagonist irbesartan in patients with systolic heart failure: a randomized double-blinded placebo-controlled study. Int J Cardiol. 2012 Nov 29;161(3):137-42. doi: 10.1016/j.ijcard.2011.07.051. PMID 21856022